CLINICAL TRIAL: NCT03408626
Title: Microbiological Assessment After Chemo-Mechanical Caries Removal Using Papain-based Enzyme Versus Conventional Rotary Tools in Occlusal Carious Lesions: Randomized Controlled Trial
Brief Title: Microbiological Assessment After Chemo-Mechanical Caries Removal Using Papain-based Enzyme Versus Conventional Rotary Tools in Occlusal Carious Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Laila Akmal Emad Eldien Elokaly, Teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBC-CU-2017-12-28
Record Dates: First submitted 2017-12-26; First posted 2018-01-24 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-07

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- papain chemomechenical caries removal agent (brix 3000) (Experimental): papain chemomechenical caries removal agent (Birx 3000) and the exclusive Encapsulating Buffer Emulsifier (EBE) technology claim it has effective and selective proteolytic action
  Interventions: Drug: Papain-based Chemo-mechanical caries removal agent; Device: conventional rotary
- conventional (Placebo Comparator): conventional 330 bur
  Interventions: Drug: Papain-based Chemo-mechanical caries removal agent; Device: conventional rotary

INTERVENTIONS:
Drug: Papain-based Chemo-mechanical caries removal agent — Birx 3000 and the exclusive Encapsulating Buffer Emulsifier (EBE) technology claim it has effective and selective proteolytic action to remove collagen fiber in the carious tissue. It has an antibacterial and antifungal power, thus it has an antiseptic power at the tissue level .furthermore, this gel does not contain chloramines in its formula, which enhances its toxicological safety feature.
  Other Names: Brix 3000
Device: conventional rotary — traditional rotary method
  Other Names: round bur 330

SUMMARY:
This study will be conducted to assess the efficacy of caries excavation using the papain-based chemo-mechanical method (Brix 3000) in comparison to conventional rotary tools in the reduction of the bacterial population in occlusal carious cavities

DETAILED DESCRIPTION:
Twenty-three patients who will fulfill the inclusion criteria will be enrolled to the study. For every patient two contra-lateral class I carious molars will be selected, so the total number of included molars will be 46 molars. One contra-lateral molar will be randomly assigned to the chemo-mechanical (Brix 3000) caries removal technique and the other will be assigned to the conventional rotary one. From every molar two dentin specimens will be collected (baseline and after excavation) with a total of 92 samples

ELIGIBILITY:
Inclusion Criteria:

1. Class I carious lesions
2. Lower molars
3. Bilateral lesions
4. 18 -50 years
5. Males or Females (Both genders)
6. Good oral hygiene
7. Co-operative patients approving the trial

Exclusion Criteria:

1. Pregnancy
2. Systemic disease or severe medical complications
3. Periodontal problem
4. Mobile teeth, arrest caries and non-vital teeth
5. Smokers
6. Xerostomia
7. Lack of compliance
8. Not received antibiotic therapy since 1 month before sampling

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
bacterial count by Digital Colony Counter | at the same visit (20 minutes)
  The number of colonies will be expressed as colony-forming units (CFU/ml) compared before and after removal caries using brix 3000 or rotary method